CLINICAL TRIAL: NCT04026035
Title: PCR Technic Evaluation in the Microbial Diagnostic of Septicemia in Hemodialysis Patients With Catheter.
Acronym: PCRDial
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Aquitaine Microbiologie (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2019/01
Record Dates: First submitted 2019-07-16; First posted 2019-07-19 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Septicemia in Hemodialysis
Keywords: PCR; hemoculture; septicemia
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aims of this study are to evaluate the PCR on whole blood approach to determine rapidly both the susceptibility and the identification of Staphylococcus responsible of septicemia in patients under hemodialysis with catheter. The results obtained with this novel experimental approach will be compared to those obtained on the same clinical samples by the routine diagnostic laboratory.

DETAILED DESCRIPTION:
The outlook of current trends indicates that maximum effort is needed to tailor the initial antimicrobial therapy in patients under hemodialysis with catheter. Specific emphasis is put on early availability of antimicrobial susceptibility results by Diagnostic laboratories to optimize the management of those difficult infections.

Direct whole blood PCR could allow a rapid determination of bacterial susceptibility to antibiotics. The study is designed to assess the concordance of a direct whole blood PCR targeting staphylococcus and its susceptibility to oracillin with the classical microbiological approach of samples from hemodialysis patients with catheter suspected of septicemia. This innovative approach should allow a faster diagnostic allowing the clinicians to better tailor the initial empirical antimicrobial therapy which has been proven crucial for a good clinical management of the patients.

Moreover, the use of an adequate antimicrobial therapy early in the management of the patients, should not only lead to a better clinical outcome but also avoid unnecessary prescriptions of drugs which are the main drivers of the emergence and spread of antimicrobial resistance.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 year old,
* suspicion of septicemia in hemodialysis patient with catheter,
* patient oral consent prior to inclusion in the study.

Exclusion Criteria:

* patients who went through the A&E department,
* patients who have received an antimicrobial therapy more than 8 hours long,
* patient under legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are treated in hemodialysis in the Nephrology Transplantation Dialysis Department of the Pellegrin Hospital of Bordeaux University Hospital. The hemodialysis unit of this service, supports a constant cohort of dialysis patients three times a week (Monday / Wednesday / Friday or Tuesday / Thursday / Saturday).
  Sepsis can occur during a hemodialysis session or be the cause of hospitalization.
  During an infectious episode, the patient is informed orally of the study and gives his oral and written consent to take an additional tube in order to carry out a bacteriological complementary analysis using a new technique to compare it to the "gold standard".
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Estimate the bacterial species concordance between the diagnostic laboratory approach and the novel approach | 48 hours after inclusion visit
  The bacterial contamination will be estimated by the results of hemoculture compared to the PCR approach. The concordance between the two profils will be observed.

SECONDARY OUTCOMES:
Evaluate the concordance of meticillin resistance diagnosis between PCR and blood cultures | 48 hours after inclusion visit
  The meticillin resistance diagnosis will be estimated by the result of PCR approach and blood cultures in hemodialysis patients with renal insufficiency with a suspected sepsis.

CONTACTS AND LOCATIONS:
Overall Officials: Fatima M'ZALI, Dr, Study Chair — Aquitaine Microbiologie
Locations (1):
- Hôpital Pellegrin - service de néphrologie, transplantation, dialyse et aphérèses, Bordeaux, France